CLINICAL TRIAL: NCT01082575
Title: Oxygen Saturation Monitoring in the General Care Floor (GCF): An Observational Study of Repetitive Reductions in Airflow
Brief Title: Oxygen Monitoring of Patients After Surgery on the Hospital General Care Floor
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COV-MO-PO-A109
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Disordered Breathing
Keywords: Post Op Patients; Continuous Pulse Oximetry Monitoring; Major Surgery
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major Surgery: Oxygen Monitoring
  Interventions: Device: Oxygen Monitoring

INTERVENTIONS:
Device: Oxygen Monitoring — No intervention
  Other Names: Nellcor Pulse Oximeter; N600X

SUMMARY:
The pain medication given after major surgery may cause some patients to stop breathing for periods of time especially at night time. An oxygen monitor may reflect this abnormal breathing pattern. This is an observational study of 100 post-operative patients who will be monitored with a pulse oximeter for a minimum of two nights and a maximum of five nights to determine the prevalence of this abnormal breathing pattern.

DETAILED DESCRIPTION:
No further details necessary or available.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Discharge from the post-anesthesia care unit (PACU) to the GCF after any of the following major surgeries: bariatric surgery, major orthopedic surgery (e.g., total hip replacement), major general surgery (e.g., bowel resections, open cholecystectomy), and major gynecological surgery (e.g., radical hysterectomy)

Exclusion Criteria:

* Pre-existing central neurological disease, including but not limited to recent traumatic brain injury, stroke, and neurodegenerative disease
* Ongoing use of mechanical ventilation or continuous positive airway pressure in the GCF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Mecca, MD, Study Chair — Medtronic - MITG
Locations (3):
- United States (3):
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Tulane University, New Orleans, Louisiana
  - Texas Health Research & Education Institute, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from February 12, 2010 to June 25, 2010 from an acute care hospital.
Pre-assignment Details: All enrolled patients were included into the trial. This was an observational study.
Groups:
- Major Surgery: Post Operative patients
Period: Overall Study
Arm/Group | Major Surgery
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Major Surgery
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.79 (12.018)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Adverse Events (AE) Caused by no Breathing
Description: Number of participants with Airway Obstruction that caused the patient to stop breathing Number of participants with Cardiac arrest w/resuscitation caused by the patient not breathing
Time Frame: Five Nights
Population: All enrolled patients
Measure: Number; unit: participants
Groups:
- General Care Floor: Observational General Care Floor Group
Arm/Group | General Care Floor
Number analyzed (Participants) | 100
participants | 0

2. Primary Outcome: Number of General Care Floor Patients Exhibiting a Saturation Pattern Detection (SPD) Alert.
Description: Number of patients on the General care Floor in which a SPD (Saturation Pattern Detection) Alert occurs. Each patient wore a sensor on their finger continuously after surgery for up to 5 days. The sensor was attached to a Nellcor N600X oximeter which measures blood oxygen level. A SPD alert detects a patient's blood oxygen level that is increasing and decreasing in a pattern that is associated with periods of no breathing.
Time Frame: 5 days
Population: 93 evaluable patients out of 100 enrolled.
Measure: Number; unit: participants
Arm/Group | General Care Floor
Number analyzed (Participants) | 93
participants | 74

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Major Surgery
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No